CLINICAL TRIAL: NCT01475032
Title: A Phase III, 12-week, Multicentre, Multinational, Randomised, Double-blind, Double-dummy, 3 Arm-parallel Group Study to Test the Efficacy of CHF 1535 (Fixed Combination of Beclomethasone Dipropionate (BDP) Plus Formoterol Fumarate (FF)) Versus a Free Combination of Beclomethasone Dipropionate Plus Formoterol Fumarate and Versus a Monotherapy of Beclomethasone Dipropionate in Partly Controlled Asthmatic Children
Brief Title: Efficacy Study of the Product "CHF 1535" Versus Beclomethasone (BDP) and Free Combo in Asthmatic Children
Acronym: PAED2/FRESH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0807-PR-0024; 2009-016757-18 (EudraCT Number)
Record Dates: First submitted 2011-10-11; First posted 2011-11-21 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; children; chronic treatment
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; alpha-ketoisovalerate dehydrogenase phosphatase; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CHF 1535 (Experimental): CHF 1535 (BDP/FF) for 12 weeks
  Interventions: Drug: CHF 1535
- BDP (Active Comparator): BDP for 12 weeks
  Interventions: Drug: Beclomethasone (BDP)
- BDP+FF (Active Comparator): free combo BDP+FF for 12 weeks
  Interventions: Drug: Beclomethasone (BDP) + Formoterol Fumarate (FF)

INTERVENTIONS:
Drug: CHF 1535 — CHF 1535 (BDP/FF) for 12 weeks
  Arms: CHF 1535
Drug: Beclomethasone (BDP) — Beclomethasone (BDP) for 12 weeks
  Arms: BDP
Drug: Beclomethasone (BDP) + Formoterol Fumarate (FF) — free combo Beclomethasone (BDP) + FF for 12 weeks
  Arms: BDP+FF

SUMMARY:
The purpose of this study is to demonstrate that CHF 1535 in pressurized metered dose inhaler (pMDI) is non-inferior to the corresponding dose of free combination of Beclomethasone (BDP) and Formoterol Fumarate (FF) and superior to the corresponding dose of BDP in terms of lung functions in asthmatic children patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children (aged ≥ 5 and < 12 years)
* Partly controlled asthma children according to Global Initiative for Asthma guidelines (GINA)
* Symptomatic asthmatic patients treated with BDP up to 400 micrograms or equivalent
* FEV1 ≥ 60% and ≤ 95% of predicted normal values

Exclusion Criteria:

* Patients with two or more admissions to hospital for asthma exacerbation in the past 12 months or any admission to intensive care ever.
* Occurrence of acute asthma exacerbations or lower respiratory tract infections in the 4 weeks before study entry
* History of near fatal asthma
* History of cystic fibrosis, bronchiectasis or primary ciliary dyskinesia
* Diagnosis of restrictive lung disease.
* Patients treated with systemic corticosteroids
* Significant medical history and/or treatments

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 638 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
pre-dose FEV1 (forced expiratory volume in the first second) | 12 weeks
  Assessment of lung function parameter as pre-dose FEV1

SECONDARY OUTCOMES:
Patient with Asthma symptoms | 12 weeks
  Patients with Asthma symptoms
FVC (forced vital capacity) | 12 weeks
  Assessment of lung function parameter as FVC
Rescue medication use | 12 weeks
  rescue medication used by the patient
PEF (peak expiratory flow) | 12 weeks
  Assessment of PEF as lung function parameter
Number of patients with adverse events | 12 weeks
  number of adverse event per patient
Blood parameters | at week 0 and week 12
  Assessment of standard blood parameters (Hematology and chemistry)
Heart rate | 12 weeks
  Assessment of heart rate
Blood pressure | 12 weeks
  Assessment of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio BARALDI, MD, Principal Investigator — University of Padova - Italy
Locations (11):
- UMHAT "Alexandrovska, Plovdiv, Bulgaria
- Necker Enfants Malades Hospital, Paris, France
- Drez. Gelb & Knecht, Bretten, Germany
- Micro Care Kft, Szigetvár, Hungary
- G.Gaslini Institute, Genoa, Italy
- Uniwersytetu Medycznego, Lodz, Poland
- Spitalul Clinic Universitar de Urgenta Elias, Bucharest, Romania
- Moscow State Medical University, Moscow, Russia
- NZZ- Detská pneumologická a ftizeologická ambulanci, Dolný Smokovec, Slovakia
- Hospital de Sabadell, Barcelona, Spain
- Institute of Pediatrics, Kyiv, Ukraine

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-016757-18